CLINICAL TRIAL: NCT05239065
Title: Knowledge Translation of Personalized Stress Management in Occupational Populations With Application of HUAWEI Portable Devices
Brief Title: Personalized Stress Management With Application of Portable Devices in Occupational Populations
Acronym: PSMPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huazhong University of Science and Technology (Other)
Collaborators: Wuhan No.1 Hospital (Other)
Responsible Party: Principal Investigator, Wei Wang, Professor, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HWTJ2019085075
Record Dates: First submitted 2021-12-13; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Stress, Psychological; Autonomic Nervous System Diseases; Emotional Stress
Keywords: Stress at work; Stress management; Autonomic system; Physical exercise; Relaxation; Knowledge translation
MeSH Terms: conditions — Stress, Psychological; Autonomic Nervous System Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized stress management nursing coaching with application of portable device (Experimental): Arm (Tongji Hospital) All the participants will receive a paper-printed brochure introducing stress and stress management strategies and the instruction of using HUAWEI portable device at the recruitment. During the 3-month intervention phase, multiple formats of stress and stress management knowledge educations will be sent by the health educator on weekly basis. The participants will have personalized stress management nursing coaching and assistance of building up new life habits, they will be also encouraged to submit a weekly questionnaire for self-evaluation. Finally, participants from Tongji hospital will be involved in a social network to share their experience anonymously and gain knowledge from the group chat.
  Interventions: Behavioral: The personalized interventions
- Minimum information transfer and assistance of building up healthy life habits (Sham Comparator): Arm2 (Wuhan No1 Hospital) - The participants will only receive a paper-printed brochure introducing stress and stress management strategies and the instruction of using HUAWEI portable device at the recruitment. There is no recurrent knowledge education, interpersonal communications, data feedbacks with the participants during the 3-month intervention phase.
  Interventions: Behavioral: The basic intervention

INTERVENTIONS:
Behavioral: The basic intervention — The participants will receive a paper-printed booklet introducing stress and stress management strategies, regular exercise, deep breathing and mediation, etc, as well as a HUAWEI portable device at the recruitment. During the following 3-month intervention phase, there is not informational materials, portable device data feedback, online group discussion or interpersonal communications with the participants. The participants will only need to fill in a simplified questionnaire biweekly.
  Arms: Minimum information transfer and assistance of building up healthy life habits
Behavioral: The personalized interventions — The participants will receive a paper-printed booklet introducing stress and stress management strategies and a HUAWEI portable device at the recruitment. A neurologist will be the health educator to host an online group for free communications. The typical stress-relieving methods and the strategies of using portable device will be explained by providing small videos, online article links and nursing coaching in person. The health educator will give regular knowledge educations about the stress hazards, stress management necessities and skills on weekly basis. The weekly data of HUAWEI portable devices will be sent to the participants along with personalized suggestions by trained nurses. At certain occasions, gifts and rewards will be sent out for encouragement and keeping attachment to the program. The participants will be required to fill in the weekly questionnaires online for feedback.
  Arms: Personalized stress management nursing coaching with application of portable device

SUMMARY:
Hospital setting is a stressful environment to the hospital staff due to work shifts, high level of responsibility, stressful challenging situations, as well as work and emotional pressures. The rate of burnout among hospital staff is high, as well as the risk of depression and suicide. The association between chronic work stress in hospital and the development of metabolic syndrome, cardiovascular complications and cancer is well established. However, it is actually not easy for the hospital staff to establish a healthier life habit and stress management skills by themselves due to the busy work schedule and the lack of persistence of building up new habits. We hypothesized that conduction of the personalized stress management coaching with the assistance of portable device could be beneficial for the hospital staff to adopt a few healthy behaviors for daily practice, which could reduce stress and the related consequences. The current study will be conducted in two separate hospitals from Wuhan (China) with different intervention strategies and conduction teams. Each institution will recruit 200 participants and complete the full set of biographic information collections at recruitment. Clinical score evaluations, biosample collections as well as 24 h Holter monitoring will be both collected at the recruitment and after 3-month intervention phase. Tongji hospital will receive the active stress-management intervention; the health educator will group the participants together and provide on a weekly basis: stress knowledge and stress-related hazards online, stress management necessities and skills. Meanwhile, weekly data of exercises, cardiac health and sleep condition generated from HUAWEI portable devices will be summarized and sent to the participants together with personalized suggestions and encouragement by trained nurses. Participants from Tongji hospital will be involved in a social network to share their experience and gain insight from the discussions. Finally, they will also complete an electronic diary that covers elements of daily life and stress management activity. The Control institution will be Wuhan No1 hospital, the participants will receive minimum information regarding stress and stress management; they will not receive personalized intervention and will not be involved in group chat. They will be asked to fill in a simplified questionnaire biweekly. The outcome parameters will be the stress relief evaluated by clinical forms and questionnaires, heart rate variability (HRV) parameters, and the establishments of healthier life habits. The current study design would propose a novel strategic stress management plan for the hospital administrates in order to improve the hospital staff health.

ELIGIBILITY:
Inclusion Criteria:

* Working as night-shift staff in Tongji hospital
* Need to keep this position for at least 6 months (no plan to leave)
* Selection will ensure a good balance of age and gender
* Willing to participate in the study and sign the consent form

Exclusion Criteria:

* Planning to leave the hospital or the units for any reason
* Not a good medical condition or context for reliable follow-up
* Having a serious medical condition (for instance cancer, stroke)
* Living in a special life context that is source of stress

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the frequency of applications of stress-relieving strategies compared to the baseline | Baseline (The first week of participating the program) , endpoint time point (The last week of participating the program), and every week between these 2 time points during the 3-month intervention
  The frequency of applications of stress-relieving strategies, including daily physical activity, deep slow breathing activity, relaxation or mindfulness meditation, which would be conducted by the participants voluntarily, will be summarized on weekly basis.
Change of the Chinese version of Perceived Stress Scale (PSS score) for evaluation of stress compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  Perceived Stress Scale (PSS score) assess the extent of feeling of nervousness and loss of control, including 14 questions. For each question, "1" for "Never", "2" for "Once in a while", "3" for "Sometimes", "4" for "Often", "5" for "Always". The total score is between 14-70.A higher score indicates a higher level of perceived stress.
Change of depression Anxiety Stress Scale (DASS score) for assessing stress, depression and anxiety compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  The Depression Anxiety Stress Scale (DASS-12) has been demonstrated to be a reliable and valid measure in assessing mental health in the Chinese population. Questions 3, 5, 10, 13, 16, 17 and 21 formed the depression subscale. The total depression subscale score was divided into normal (0-9), mild depression (10-12), moderate depression (13-20), severe depression (21-27), and extremely severe depression (28-42). Questions 2, 4, 7, 9, 15, 19, and 20 formed the anxiety subscale. The total anxiety subscale score was divided into normal (0-6), mild anxiety (7-9), moderate anxiety (10-14), severe anxiety (15-19), and extremely severe anxiety (20-42). Questions 1, 6, 8, 11, 12, 14, and 18 formed the stress subscale. The total stress subscale score was divided into normal (0-10), mild stress (11-18), moderate stress (19-26), severe stress (27-34), and extremely severe stress (35-42).
Change of trier work-stress scale (TICS-9 scale) for evaluating the sources of chronic stress in daily life compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  The Trier Inventory for Chronic Stress (TICS) is a standardized questionnaire for assessing nine interrelated factors of chronic stress from 9 dimensions: Work Overload, Social Overload, Pressure to Perform, Work Discontent, Excessive Demands from Work, Lack of Social Recognition, Social Tensions, Social Isolation, and Chronic Worrying. The TICS-9 is a short version of the original 57-item TICS. This version includes nine items reflecting all dimensions of the long version. The items can be rated from 0 to 5 (0 = never, 1 = rarely, 2 = sometimes, 3 = often, 4 = very often). Higher values suggest greater stress. Satisfactory psychometrics have been evidenced in several studies, with Cronbach's Alpha ranging from α = 0.88-0.91.
Change of the Fatigue Scale (FAS) for evaluating fatigue compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  The Fatigue Scale (FAS) was used to measure total fatigue, and includes 10 items rated on a 5-point rating scale (1=never~ 5=always). This scale has good reliability and content validity for measuring fatigue in a general or worker population.
Change of the Epworth Sleepiness Scale for sleep quality compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  The Epworth Sleepiness Scale (ESS) includes 8 items and assesses the general level of daytime sleepiness. Scores range from 0-24 where higher scores indicate greater sleepiness. Following the developer's suggestion, a score greater than 10 was classified as high daytime sleepiness.
Change of the Subjective Happiness Scale (SHS) for evaluating subjective global happiness compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  The Subjective Happiness Scale (SHS) is a four-item measure of subjective global happiness rated on a seven-point Likert scale. A single SHS score is the mean of the responses to the four items. SHS scores can range from 1 to 7, where a higher score indicates a higher level of happiness.
Change of heart rate variability (HRV) parameters (time-domain analysis:SDNN, SDNN index, SDANN index, RMMSD) for assessing the autonomic nervous system compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  Heart rate variability (HRV) to assess the autonomic nervous system using different parameters from time-domain analysis (SDNN, SDNN index, SDANN index, RMMSD), the unit for these parameters are all "millisecond". The participants will have 24 hr cardiac holter monitoring at the recruitment and the last day of 3-month intervention.
  SDNN: Standard deviation of NN intervals, NN interval is the time (normalized) between two detected heartbeat detections. (unit: ms) SDANN: Standard deviation of the average NN intervals for each 5 min segment of a 24 h HRV recording. (unit: ms) SDNN index: Mean of the standard deviations of all the NN intervals for each 5 min segment of a 24 h HRV recording. (unit: ms) RMMSD: Root mean square of successive RR interval differences. (unit: ms)
Change of heart rate variability (HRV) parameters (time-domain analysis: pNN50) for assessing the autonomic nervous system compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  Heart rate variability (HRV) to assess the autonomic nervous system using different parameters from time-domain analysis (pNN50), the unit for these parameters are all "percentage %". The participants will have 24 hr cardiac holter monitoring at the recruitment and the last day of 3-month intervention.
  pNN50: Percentage of successive RR intervals that differ by more than 50 ms. (unit: %)
Change of heart rate variability (HRV) parameters (frequency-domain analysis: VLF power, LF power, HF power) for assessing the autonomic nervous system compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  Heart rate variability (HRV) to assess the autonomic nervous system using different parameters from frequency-domain analysis (VLF power, LF power, HF power), all the units are "ms2". The participants will have 24 hr cardiac holter monitoring at the recruitment and the last day of 3-month intervention.
  VLF (very-low-frequency) power: Absolute power of the very-low-frequency band (0.0033-0.04 Hz) (unit: ms2).
  LF (low-frequency) power: Absolute power of the low-frequency band (0.04-0.15 Hz)(unit: ms2).
  HF (high-frequency) power: Absolute power of the high-frequency band (0.15-0.4 Hz) (unit: ms2).
Change of heart rate variability (HRV) parameters (frequency-domain analysis: LF/HF) for assessing the autonomic nervous system compared to the baseline | Baseline (at recruitment) and endpoint (the last day of 3-month intervention)
  Heart rate variability (HRV) to assess the autonomic nervous system using different parameters from frequency-domain analysis (LF/HF), the unit is "percentage %". The participants will have 24 hr cardiac holter monitoring at the recruitment and the last day of 3-month intervention.
  LF/HF: Ratio of LF(low-frequency)-to-HF(high-frequency) power.(unit: %).

SECONDARY OUTCOMES:
Change of the daily travel distance as evaluated by portable device compared to the baseline | Daily during the 3-month intervention (during the time of wearing the HUAWEI bracelet)
  The participants will be encouraged to wear HUAWEI bracelet on daily basis to monitor the amount of exercise. The daily travel distance recorded by the bracelet will be summarized to reveal the difference along with the time of interventions.
Change of medium-to-high level exercise time duration as evaluated by portable device compared to the baseline | Daily during the 3-month intervention (during the time of wearing the HUAWEI bracelet)
  The participants will be encouraged to wear HUAWEI bracelet on daily basis to monitor the amount of exercise. The time duration of conducting medium-to-high level exercise recorded by the bracelet will be summarized to reveal the difference along with the time of interventions.
Change of the total steps traveled daily as evaluated by portable device compared to the baseline | Daily during the 3-month intervention (during the time of wearing the HUAWEI bracelet)
  The participants will be encouraged to wear HUAWEI bracelet on daily basis to monitor the amount of exercise. The total steps traveled daily recorded by the bracelet will be summarized to reveal the difference along with the time of interventions.
Change of the daily duration for wearing portable device compared to the baseline | Daily during the 3-month intervention (during the time of wearing the HUAWEI bracelet)
  The participants will be encouraged to wear HUAWEI bracelet on daily basis. The daily duration for wearing HUAWEI bracelet will be summarized to reveal the difference along with the time of interventions to reflect the establishment of the habit of wearing portable device.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dziembowska I, Izdebski P, Rasmus A, Brudny J, Grzelczak M, Cysewski P. Effects of Heart Rate Variability Biofeedback on EEG Alpha Asymmetry and Anxiety Symptoms in Male Athletes: A Pilot Study. Appl Psychophysiol Biofeedback. 2016 Jun;41(2):141-50. doi: 10.1007/s10484-015-9319-4. PMID 26459346
- [Background] Scherz WD, Seepold R, Madrid NM, Crippa P, Ortega JA. RR interval analysis for the distinction between stress, physical activity and no activity using a portable ECG. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:4522-4526. doi: 10.1109/EMBC44109.2020.9175458. PMID 33018999
- [Result] Harvey SB, Epstein RM, Glozier N, Petrie K, Strudwick J, Gayed A, Dean K, Henderson M. Mental illness and suicide among physicians. Lancet. 2021 Sep 4;398(10303):920-930. doi: 10.1016/S0140-6736(21)01596-8. PMID 34481571
- [Result] Marchalik D. Physician burnout in the modern era. Lancet. 2019 Mar 2;393(10174):868-869. doi: 10.1016/S0140-6736(19)30399-X. No abstract available. PMID 30837137
- [Result] West CP, Dyrbye LN, Erwin PJ, Shanafelt TD. Interventions to prevent and reduce physician burnout: a systematic review and meta-analysis. Lancet. 2016 Nov 5;388(10057):2272-2281. doi: 10.1016/S0140-6736(16)31279-X. Epub 2016 Sep 28. PMID 27692469
- [Result] Debnath S, Levy TJ, Bellehsen M, Schwartz RM, Barnaby DP, Zanos S, Volpe BT, Zanos TP. A method to quantify autonomic nervous system function in healthy, able-bodied individuals. Bioelectron Med. 2021 Aug 27;7(1):13. doi: 10.1186/s42234-021-00075-7. PMID 34446089
- [Result] Hamasaki H. Effects of Diaphragmatic Breathing on Health: A Narrative Review. Medicines (Basel). 2020 Oct 15;7(10):65. doi: 10.3390/medicines7100065. PMID 33076360
- [Result] De Couck M, Caers R, Musch L, Fliegauf J, Giangreco A, Gidron Y. How breathing can help you make better decisions: Two studies on the effects of breathing patterns on heart rate variability and decision-making in business cases. Int J Psychophysiol. 2019 May;139:1-9. doi: 10.1016/j.ijpsycho.2019.02.011. Epub 2019 Mar 1. PMID 30826382
- [Result] Davila MI, Lewis GF, Porges SW. The PhysioCam: A Novel Non-Contact Sensor to Measure Heart Rate Variability in Clinical and Field Applications. Front Public Health. 2017 Nov 22;5:300. doi: 10.3389/fpubh.2017.00300. eCollection 2017. PMID 29214150
- [Result] Bonaz B, Sinniger V, Pellissier S. Vagal tone: effects on sensitivity, motility, and inflammation. Neurogastroenterol Motil. 2016 Apr;28(4):455-62. doi: 10.1111/nmo.12817. PMID 27010234
- [Result] Prinsloo GE, Derman WE, Lambert MI, Laurie Rauch HG. The effect of a single session of short duration biofeedback-induced deep breathing on measures of heart rate variability during laboratory-induced cognitive stress: a pilot study. Appl Psychophysiol Biofeedback. 2013 Jun;38(2):81-90. doi: 10.1007/s10484-013-9210-0. PMID 23435801
- [Result] Aguilar-Raab C, Stoffel M, Hernandez C, Rahn S, Moessner M, Steinhilber B, Ditzen B. Effects of a mindfulness-based intervention on mindfulness, stress, salivary alpha-amylase and cortisol in everyday life. Psychophysiology. 2021 Dec;58(12):e13937. doi: 10.1111/psyp.13937. Epub 2021 Sep 15. PMID 34525214
- [Result] Watford TS, O'Brien WH, Koerten HR, Bogusch LM, Moeller MT, Sonia Singh R, Sims TE. The mindful attention and awareness scale is associated with lower levels of high-frequency heart rate variability in a laboratory context. Psychophysiology. 2020 Mar;57(3):e13506. doi: 10.1111/psyp.13506. Epub 2019 Nov 17. PMID 31737916
- [Result] Chin MS, Kales SN. Understanding mind-body disciplines: A pilot study of paced breathing and dynamic muscle contraction on autonomic nervous system reactivity. Stress Health. 2019 Oct;35(4):542-548. doi: 10.1002/smi.2887. Epub 2019 Sep 5. PMID 31347763
- [Result] Reive C. The Biological Measurements of Mindfulness-based Stress Reduction: A Systematic Review. Explore (NY). 2019 Jul-Aug;15(4):295-307. doi: 10.1016/j.explore.2019.01.001. Epub 2019 Jan 18. PMID 30765300
- [Result] Heckenberg RA, Eddy P, Kent S, Wright BJ. Do workplace-based mindfulness meditation programs improve physiological indices of stress? A systematic review and meta-analysis. J Psychosom Res. 2018 Nov;114:62-71. doi: 10.1016/j.jpsychores.2018.09.010. Epub 2018 Sep 22. PMID 30314581
- [Result] Park C. Mind-body CAM interventions: current status and considerations for integration into clinical health psychology. J Clin Psychol. 2013 Jan;69(1):45-63. doi: 10.1002/jclp.21910. Epub 2012 Aug 30. PMID 22936306
- [Result] Rathbone AL, Prescott J. The Use of Mobile Apps and SMS Messaging as Physical and Mental Health Interventions: Systematic Review. J Med Internet Res. 2017 Aug 24;19(8):e295. doi: 10.2196/jmir.7740. PMID 28838887
- [Result] Lemaire JB, Wallace JE, Lewin AM, de Grood J, Schaefer JP. The effect of a biofeedback-based stress management tool on physician stress: a randomized controlled clinical trial. Open Med. 2011;5(4):e154-63. Epub 2011 Oct 4. PMID 22567069
- [Result] Malmberg Gavelin H, Eskilsson T, Boraxbekk CJ, Josefsson M, Stigsdotter Neely A, Slunga Jarvholm L. Rehabilitation for improved cognition in patients with stress-related exhaustion disorder: RECO - a randomized clinical trial. Stress. 2018 Jul;21(4):279-291. doi: 10.1080/10253890.2018.1461833. Epub 2018 Apr 25. PMID 29693483
- [Derived] Liu W, Wang Q, Zheng D, Mei J, Lu J, Chen G, Wang W, Ding F. The Effects of a Complex Interactive Multimodal Intervention on Personalized Stress Management Among Health Care Workers in China: Nonrandomized Controlled Study. J Med Internet Res. 2024 Jul 12;26:e45422. doi: 10.2196/45422. PMID 38996333
- [Derived] Wang Q, Collet JP, Mei J, Chen G, Huang S, Yang Y, Wang W, Ding F. Complex interactive multimodal intervention to improve personalized stress management among healthcare workers in China: A knowledge translation protocol. Digit Health. 2023 Jul 24;9:20552076231184052. doi: 10.1177/20552076231184052. eCollection 2023 Jan-Dec. PMID 37545629